CLINICAL TRIAL: NCT03252795
Title: Uterus Transplantation From a Multi-organ Donor: A Prospective Trial
Brief Title: Uterus Transplantation From a Multi-organ Donor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2016/0731
Record Dates: First submitted 2017-06-22; First posted 2017-08-17 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Mayer Rokitansky Kuster Hauser Syndrome
Keywords: Infertility, female; Mayer Rokitansky Kuster Hauser Syndrome; Transplantation; Deceased donor
MeSH Terms: conditions — Infertility, Female; Mullerian aplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterus transplantation (Experimental)
  Interventions: Procedure: uterus transplantation

INTERVENTIONS:
Procedure: uterus transplantation — transplantation of a uterus from a deceased donor

SUMMARY:
Uterus transplantation: screening, in vitro fertilization [IVF] treatment to be able to freeze embryos, uterus transplantation, pregnancy and afterwards removal of the uterus.

ELIGIBILITY:
Inclusion Criteria:

* Female with Maier-Rokitansky-Kuster-Hauser syndrome
* Mucosal neovagina of at least 7 cm
* In a stable relationship for at least 1 year
* Child wish
* Good renal function (and presence of both kidneys)
* Psychologically stable and compliant
* At least 8 frozen embryos after IVF/intracytoplasmic sperm injection [ICSI]
* Living in Belgium and a good health insurance
* Willing and able to provide informed consent

Exclusion Criteria:

* Major pelvic surgery
* Major chronic illnesses
* Other risk factors or malignancies
* BMI > 30

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival of the uterus 1 year after transplantation | 1 year after uterus transplantation
  Survival of the uterus 1 year after transplantation
Complications after uterus transplantation | As long as the uterus remains in situ (the uterus will be removed within one year after delivery)
  Complications after uterus transplantation
Ongoing pregnancy rate | 4 weeks after embryo transfer
  Ongoing pregnancy rate
Take home baby rate | 9 months after embryo transfer
  Take home baby rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital - Women's Clinic, Ghent, Belgium